CLINICAL TRIAL: NCT05288881
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Intravenous ANX105 in Normal Healthy Volunteers
Brief Title: Single Ascending Dose Study of ANX105
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Annexon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ANX105-NHV-01; 2021-005510-33 (EudraCT Number)
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Healthy

STUDY DESIGN:
Intervention Model Description: Placebo-controlled single ascending dose study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ANX105 (Experimental)
  Interventions: Biological: ANX105
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: ANX105 — Participants will receive single-ascending doses of ANX105 administered by IV infusion.
  Arms: ANX105
Drug: Placebo — Participants will receive matching placebo administered by IV infusion.
  Arms: Placebo

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of single ascending doses of ANX105 administered intravenously (IV) to healthy participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, and laboratory tests.
* Have been fully vaccinated with SARS-CoV-2 vaccination according to local guidelines within 14 days prior to Day -1.
* Documented history of vaccinations within 5 years or willing to undergo vaccinations prior to screening visit against encapsulated bacterial pathogens.

Key Exclusion Criteria:

* Clinically significant infection within 30 days prior to Day -1 that required medical intervention.
* Significant allergies to humanized monoclonal antibodies.
* Use of immunosuppressants including high-dose systemic corticosteroids within 30 days prior to Day -1.
* Antinuclear antibodies (ANA) titer ≥1:160 (for either of the 2 ANA results a minimum of 2 weeks apart) at Screening.
* Have poor venous access limiting phlebotomy.
* Donation or loss of > 500 milliliter whole blood within 30 days prior to Day 1 or donation of plasma within 14 days prior to Day -1.
* Hospitalization during the 4 weeks prior to Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2023-06-19 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Experienced Treatment-Emergent Adverse Events | Up to Week 7

SECONDARY OUTCOMES:
Amount of Serum Total Hemolytic Complement (CH50) | Up to Week 7
  Blood samples will be obtained to determine the amount of CH50.
Change from Baseline in Amount of Unbound Complement 1q (C1q) in Serum | Baseline, Week 7
  Blood samples will be obtained to determine the amount of C1q.
Amount of C1q in Cerebrospinal fluid (CSF) | Up to Week 7
  CSF samples will be obtained to determine the amount of C1q.
Serum Concentrations of ANX105 | Up to Week 7
  Blood samples will be obtained to determine serum concentrations of ANX105.
Maximum Observed Serum Concentration (Cmax) of ANX105 | Up to Week 7
  Blood samples will be obtained to determine the Cmax of ANX105.
Area Under the ANX105 Serum Concentration-Time Curve (AUC) | Up to Week 7
  Blood samples will be obtained to determine the AUC of ANX105.
CSF Concentrations of ANX105 | Up to Week 7
  CSF samples will be obtained to determine CSF concentrations of ANX105.

CONTACTS AND LOCATIONS:
Overall Officials: Olga Bandman, MD, Study Director — Annexon, Inc.
Locations (2):
- Netherlands (2):
  - Annexon Investigational Site 02, Groningen
  - Annexon Investigational Site 01, Leiden

IPD SHARING:
Plan to Share IPD: No